CLINICAL TRIAL: NCT03111537
Title: Project 4: Clinical Trial Method for Assessing a Tobacco Product Part of Models for Tobacco Product Evaluation:
Brief Title: Methods Project 4: Clinical Trial - Amended
Acronym: COMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2012NTLS050b
Record Dates: First submitted 2015-05-21; First posted 2017-04-13 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Tobacco Smoking
Keywords: cigarette; smoking; e-cigarette; nicotine replacement therapy; nrt; tobacco
MeSH Terms: conditions — Tobacco Smoking; Smoking; Vaping | interventions — Tobacco Products; Electronic Nicotine Delivery Systems; Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual Brand Cigarette (Experimental): Smoking usual brand cigarette controls, who after 8-weeks will be offered alternative nicotine products and instructed for partial or complete substitution of cigarettes (subject's choice);
  Interventions: Other: Cigarettes
- Complete Substitution E-Cigarette (Experimental): Complete substitution (i.e., no smoking) with e-cigarette use
  Interventions: Other: E-Cigarette
- Partial Substitution E-Cigarette (Experimental): Partial substitution, encouraged to use e-cigarettes instead of smoking usual cigarettes
  Interventions: Other: Cigarettes; Other: E-Cigarette
- Complete Substitution Nic Gum or Lozenge (Experimental): Complete substitution (i.e., no smoking) to nicotine gum or lozenge use
  Interventions: Other: Nicotine Gum or Lozenge

INTERVENTIONS:
Other: Cigarettes — Smoke their usual brand of cigarettes and follow their normal patterns of use.
  Arms: Partial Substitution E-Cigarette; Usual Brand Cigarette
Other: E-Cigarette — Use of E-cigarette: multiple flavors offered.
  Arms: Complete Substitution E-Cigarette; Partial Substitution E-Cigarette
Other: Nicotine Gum or Lozenge — Subject choice: Use of nicotine gum or nicotine lozenge, multiple flavors offered
  Arms: Complete Substitution Nic Gum or Lozenge

SUMMARY:
Cigarette smokers will be randomized to E-cigarette, Nicotine Gum or Lozenge, or Control Group. Participants will enter a 1 week sampling phase. Smokers interested in continuing with the study after the sampling phase will undergo a 2 week baseline assessment phase and will then enter an 8 week intervention. Tobacco use patterns, subjective responses to product, and nicotine and toxicant exposure will be assessed.

DETAILED DESCRIPTION:
Sampling period (1 week): Subjects will be randomized to an alternative nicotine product (E-cigarette, Nicotine Gum or Lozenge) or assigned to continue smoking their usual brand cigarettes. Subjects will complete screening assessments, asked to sample the assigned product and start recording their cigarette or other tobacco intake on a daily basis using an interactive voice response system (IVR). Smokers assigned to the control condition (smoking usual brand cigarettes) will be asked to choose the product that they would like to sample.

Baseline smoking period: After sampling, subjects who meet specific criteria will continue with the experimental intervention phase. These subjects will be required to attend 2 baseline clinic visits where baseline assessments will be captured. Records of their cigarette or other tobacco intake on a daily basis will continue using the interactive voice response system (IVR).

Experimental Period: After the baseline assessment, subjects will be instructed to either partially or completely substitute their cigarette smoking with their assigned product. They will assigned to one of six experimental conditions:

1. smoking usual brand cigarette controls, who after 8-weeks will be offered any of the other nicotine products to use as they choose for 8 weeks;
2. complete substitution (i.e., no smoking) with an E-cigarette;
3. partial substitution with an E-cigarette;
4. complete substitution (i.e., no smoking) with nicotine gum or nicotine lozenge.

The assigned product, E-cigarette, Nic Gum or Lozenge, but not usual brand cigarettes, will be provided to subjects at the clinic visits. Subjects will attend clinic visits over the next 8 weeks where tobacco use patterns and biomarker data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are at least 18 years of age;
* Daily smoker;
* Generally good health;
* Subject has provided written informed consent to participate in the study (adolescents under the age of 18 will be excluded because this project involves continued use of tobacco products and new tobacco products);

Exclusion Criteria:

* Unstable health;
* Pregnant or breastfeeding (due to toxic effects from tobacco products);
* Unable to read for comprehension or completion of study documents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2015-05; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Compare total nicotine equivalents (TNE) based on differing instructions for oral tobacco, nicotine replacement or e-cigarette use. | 6 months
  Compare the exposure to nicotine in the two instructions for use arms (complete substitution vs. partial substitution) across study products and compared to medicinal nicotine products and usual brand cigarettes.
Determine stabilization of product use (e.g., cigarette, oral tobacco, e-cigarette or medicinal nicotine patterns of use). | 6 months
  Examining time effects for patterns of use of cigarettes, nicotine replacement, oral tobacco or e-cigarette.
Consumer perception of the product and response to the product after sampling. | 6 months
  Consumer perception of the product evidenced by choice of which product to use in the trial after sampling.
Compare NNK exposure based on differing instructions for oral tobacco, nicotine replacement or e-cigarette use. | 8 weeks
  Complete substitution vs. partial substitution of study products for cigarettes and compare the exposure to NNK by analyzing NNAL levels in subject urine. These products are compared to medicinal nicotine products and usual brand cigarettes.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Roswell Park Cancer Center, Buffalo, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio